CLINICAL TRIAL: NCT07328048
Title: Combine Effects of Senobi Exercise & Aerobic Exercises on Body Mass Index, Fatigue and Quality of Life in Polycystic Ovarian Syndrome.
Brief Title: Effects of Senobi Exercise & Aerobic Exercises in Polycystic Ovarian Syndrome
Acronym: CESAEBMIFQPCOS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Wajeeha Zia, Assistant Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Syeda Iram Shahzadi
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovarian Syndrome Females
Keywords: Senobi; females; BMI; Fatigue; Quality of life; PCOS
MeSH Terms: conditions — Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (experimental group) (Experimental): The participants in group A will receive interventional treatment (senobi exercises), 3 days a week for 6 weeks as a supervised exercise program, as well as they will receive aerobic exercises on treadmill with 10% grade and 5mph speed for 20 minutes a session with 5 minutes of warm up and 5 minutes of cool down of total 30 minutes a session, 5 sessions for a week for 6 weeks. Baseline treatment for both groups will be deep Breathing exercise- 5 reps/3 seconds inspiration 6 seconds expiration/1 set. Self-stretching exercise for biceps and triceps- 5 reps/5 seconds hold/1 set and walking for 3 alternate days per week for 6 weeks as a home exercise program.
  Interventions: Other: Senobi exercises with aerobics exercises
- Group B (control group) (Experimental): The participants in group B will receive aerobic exercises on treadmill ( fig. 2) with 10% grade and 5mph speed for 20 minutes a session with 5 minutes of warm up and 5 minutes of cool down of total 30 minutes a session, 5 sessions for a week for 6 weeks. Subjects will be assessed at baseline and after 6 weeks. The post-interventional assessment will be taken and the results will be interpreted. Baseline treatment for both groups will be deep Breathing exercise- 5 reps/3 seconds inspiration 6 seconds expiration/1 set. Self-stretching exercise for biceps and triceps- 5 reps/5 seconds hold/1 set and walking for 3 alternate days per week for 6 weeks as a home exercise program.
  Interventions: Other: aerobic exercises

INTERVENTIONS:
Other: Senobi exercises with aerobics exercises — The participants in group A will receive interventional treatment (senobi exercises), 3 days a week for 6 weeks as a supervised exercise program, as well as they will receive aerobic exercises on treadmill with 10% grade and 5mph speed for 20 minutes a session with 5 minutes of warm up and 5 minutes of cool down of total 30 minutes a session, 5 sessions for a week for 6 weeks. Baseline treatment for both groups will be deep Breathing exercise- 5 reps/3 seconds inspiration 6 seconds expiration/1 set. Self-stretching exercise for biceps and triceps- 5 reps/5 seconds hold/1 set and walking for 3 alternate days per week for 6 weeks as a home exercise program.
  Arms: Group A (experimental group)
Other: aerobic exercises — The participants in group B will receive aerobic exercises on treadmill with 10% grade and 5mph speed for 20 minutes a session with 5 minutes of warm up and 5 minutes of cool down of total 30 minutes a session, 5 sessions for a week for 6 weeks. Subjects will be assessed at baseline and after 6 weeks. The post-interventional assessment will be taken and the results will be interpreted. Baseline treatment for both groups will be deep Breathing exercise- 5 reps/3 seconds inspiration 6 seconds expiration/1 set. Self-stretching exercise for biceps and triceps- 5 reps/5 seconds hold/1 set and walking for 3 alternate days per week for 6 weeks as a home exercise program.
  Arms: Group B (control group)

SUMMARY:
One of the most prevalent endocrine system conditions affecting women of reproductive age is polycystic ovary syndrome (PCOS), also known as hyperandrogenic anovulation (HA) or Stein-Leventhal syndrome. This chronic and heterogeneous disorder manifests itself as menstrual dysfunction, infertility, hirsutism, acne, and obesity. This study will be randomized controlled trial and will be conducted in Qasim Sandhu medical complex, Iiffat Anwar Medical Complex and OMC Hospital Lahore. Data will be collected 10 months after approval of synopsis. The total duration of treatment will be 6 weeks. Non-probability convenience sampling technique will be used and 32 participants will be recruited in study after randomization according to selection criteria. The subjects will be divided into two groups, 16 participants in each group. Group A (experimental group) will receive senobi exercises and aerobic exercises, 3 days\week for 6 weeks and Group B (control group) will receive aerobic exercises, 3days\week for 6 week.

DETAILED DESCRIPTION:
One of the most prevalent endocrine system conditions affecting women of reproductive age is polycystic ovary syndrome (PCOS), also known as hyperandrogenic anovulation (HA) or Stein-Leventhal syndrome. This chronic and heterogeneous disorder manifests itself as menstrual dysfunction, infertility, hirsutism, acne, and obesity. It is usually only diagnosed when complications develop that significantly reduce a patient's quality of life (e.g., hair loss, alopecia, acne, and infertility-related problems). The World Health Organization (WHO) estimates that in 2012 PCOS affected 116 million women globally. Although PCOS can occur at any age, beginning with menarche, the majority of instances are identified between the ages of 20 and 30. Polycystic ovary syndrome (PCOS) is an important and highly prevalent obesity-related comorbidity that develops in girls and women who are genetically predisposed to its development. This study will be randomized controlled trial and will be conducted in Qasim Sandhu medical complex, Iiffat Anwar Medical Complex and OMC Hospital Lahore. Data will be collected 10 months after approval of synopsis. The total duration of treatment will be 6 weeks. Non-probability convenience sampling technique will be used and 32 participants will be recruited in study after randomization according to selection criteria. The subjects will be divided into two groups, 16 participants in each group. Group A (experimental group) will receive senobi exercises and aerobic exercises, 3 days\week for 6 weeks and Group B (control group) will receive aerobic exercises, 3days\week for 6 week. Nutritional counselling and deep breath for 5 minutes will be used as Baseline treatment. The tools that will be used are BMI Calculator for obesity, WHQOL-BREF Questionnaire for Quality of life and multidimensional fatigue inventory (MFI) questionnaire to assess fatigue. After data collection data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Women between the Ages of 18 to 35 Diagnosed with PCOS Menstrual disturbance > 3 months BMI of 29-35kg/m Unmarried and married with multiparous

Exclusion Criteria:

* Women with other causes of menstrual disturbances (ovarian cancer) Known cardiovascular problems (cardiac arrhythmias) Uncontrolled hypertension or low blood pressure Presence of neurological disease (epilepsy, autism) Orthopedic illness (rheumatoid arthritis, osteoporosis) Cardiopulmonary disease (CVD, COPD) Musculoskeletal injuries (fracture, tendon rupture) Antiobesity medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females with PCOS
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
WHQOL-BREF Questionnaire | 6 weeks
  WHOQOL-BREF questionnaire is a reliable instrument to measure quality of life. QOL-BREF (WHOQOLBREF) questionnaire which captures many subjective aspects of QOL. This questionnaire is one of the best known instruments that has been developed for cross-cultural comparisons of QOL and is available in many languages. This instrument, by focusing on individuals' own views of their well-being, provides a new perspective on life. Its internal consistency is (α = 0.925).
Multidimensional fatigue inventory | 6 weeks
  The Multidimensional Fatigue Inventory (MFI-20) is a valid tool for assessment of fatigue. MFI-20 covering general fatigue, physical fatigue, mental fatigue, reduced activity and reduced motivation has been widely used in patients with chronic fatigue syndrome. The internal consistency of MFI-20 is (Cronbach's alpha = 0.89).
Body Mass Index | 6 weeks
  Body mass index (BMI), is a measurement tool based on a person's height and weight, and allows the classification of individuals into categories such as obese or overweight. Body mass index (BMI) is one of the ways to measure obesity in the population. Body mass index (BMI) can be calculated via mathematical operations where height and weight values are used to estimate the health status of a person.

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International University, Lahore, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Motta AB. The role of obesity in the development of polycystic ovary syndrome. Curr Pharm Des. 2012;18(17):2482-91. doi: 10.2174/13816128112092482. PMID 22376149
- [Background] Barber TM, Franks S. Obesity and polycystic ovary syndrome. Clin Endocrinol (Oxf). 2021 Oct;95(4):531-541. doi: 10.1111/cen.14421. Epub 2021 Jan 31. PMID 33460482
- [Background] Norman RJ, Dewailly D, Legro RS, Hickey TE. Polycystic ovary syndrome. Lancet. 2007 Aug 25;370(9588):685-97. doi: 10.1016/S0140-6736(07)61345-2. PMID 17720020
- [Background] Merkin SS, Phy JL, Sites CK, Yang D. Environmental determinants of polycystic ovary syndrome. Fertil Steril. 2016 Jul;106(1):16-24. doi: 10.1016/j.fertnstert.2016.05.011. Epub 2016 May 27. PMID 27240194
- [Background] Lujan ME, Chizen DR, Pierson RA. Diagnostic criteria for polycystic ovary syndrome: pitfalls and controversies. J Obstet Gynaecol Can. 2008 Aug;30(8):671-679. doi: 10.1016/S1701-2163(16)32915-2. PMID 18786289
- [Background] Hashemipour M, Amini M, Iranpour R, Sadri GH, Javaheri N, Haghighi S, Hovsepian S, Javadi AA, Nematbakhsh M, Sattari G. Prevalence of congenital hypothyroidism in Isfahan, Iran: results of a survey on 20,000 neonates. Horm Res. 2004;62(2):79-83. doi: 10.1159/000079392. Epub 2004 Jun 24. PMID 15237248
- [Background] Liu J, Wu Q, Hao Y, Jiao M, Wang X, Jiang S, Han L. Measuring the global disease burden of polycystic ovary syndrome in 194 countries: Global Burden of Disease Study 2017. Hum Reprod. 2021 Mar 18;36(4):1108-1119. doi: 10.1093/humrep/deaa371. PMID 33501984
- [Background] Bremer AA. Polycystic ovary syndrome in the pediatric population. Metab Syndr Relat Disord. 2010 Oct;8(5):375-94. doi: 10.1089/met.2010.0039. PMID 20939704
- [Background] Singh S, Pal N, Shubham S, Sarma DK, Verma V, Marotta F, Kumar M. Polycystic Ovary Syndrome: Etiology, Current Management, and Future Therapeutics. J Clin Med. 2023 Feb 11;12(4):1454. doi: 10.3390/jcm12041454. PMID 36835989
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15237248/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18786289/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27240194/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17720020/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/33460482/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22376149/